CLINICAL TRIAL: NCT06515379
Title: Emergency Department Management of Patients With Renal Infarction
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RENAL INFARCTION
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Renal Infarct; Renal Infarction - Venous; Renal Infarction - Arterial
Keywords: Renal Infarction; Emergency Department
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Renal Infarction: Patients diagnosed with renal infarction using data obtained from the hospital system have been reviewed and evaluated. Laboratory, clinical and imaging data ahve been registered and statistical analyses have been conducted

SUMMARY:
The aim of this study is to investigate laboratory parameters from medical records of patients diagnosed with renal infarction in our emergency clinic to establish early diagnostic indicators. Additionally, we will evaluate imaging methods such as CT or CT angiography and identify mortality-morbidity markers to contribute to the literature.

DETAILED DESCRIPTION:
It is planned to include 80 patients who presented to the hospital emergency department and were diagnosed with renal infarction between January 1, 2014, and June 1, 2023, in the study.

he data of patients diagnosed with renal infarction will be retrospectively collected from the hospital database and recorded in a data collection form. This includes information such as CBC (complete blood count), neutrophils, lymphocytes, platelets, lactate, anion gap, pH, bicarbonate, creatinine, urea, AST, ALT, fibrinogen, D-dimer, LDH, CRP, CT scan, and CT angiography results. Patients' demographic characteristics, physical examination findings, imaging, and laboratory results will be evaluated using patient records and the hospital registry system.

Our aim is to identify early morbidity and mortality indicators in cases of renal infarction where diagnosis is often delayed or missed, contributing to the survival of patients. We believe that the findings from our statistical analysis can guide routine practice, especially in the management of patients presenting to the emergency department with complaints of abdominal and/or flank pain

ELIGIBILITY:
Inclusion criteria:

Adult patients aged 18 years and older Cases diagnosed with renal infarction presenting to the Emergency Department of Dışkapı Yıldırım Beyazıt Training and Research Hospital

Exclusion criteria:

Patients without imaging methods Patients with incomplete laboratory and file follow-ups Patients previously diagnosed with renal infarction and currently under treatment Patients diagnosed with other clinical conditions such as pyelonephritis, lower urinary tract infections, nephrolithiasis

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients administered to emergency department and diagnosed with renal infarction will be retrospectively determined from hospital data system.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Renal Infarction | 9 years
  patients diagnosed with renal infarction

CONTACTS AND LOCATIONS:
Overall Officials: gulsen akcay, ass. prof., Study Director — ass. prof. of organization
Locations (1):
- Diskapi Teaching and Research Hospital, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Delezire A, Terrasse M, Bouet J, Laot M, Brun V, Oger E, Vigneau C. Acute renal infarction: long-term renal outcome and prognostic factors. J Nephrol. 2021 Oct;34(5):1501-1509. doi: 10.1007/s40620-020-00953-4. Epub 2021 Mar 25. PMID 33765299
- [Background] Francisco D, Pimenta G, Martins AC, Laranjinha I, Estibeiro H, Gil C, Goncalves M, Gaspar MA. Recovering from a renal vascular catastrophe: Case report. Clin Nephrol Case Stud. 2023 Mar 5;11:44-49. doi: 10.5414/CNCS110984. eCollection 2023. PMID 36896140
- [Background] Woo S, Lee CA, Lee JW, Moon J, Cho YS, Nah S, Han S. Predictors for Distinguishing Renal Infarction From Urolithiasis in the Emergency Department: A Randomly Matched Retrospective Case-Control Study. J Emerg Med. 2023 Jan;64(1):31-39. doi: 10.1016/j.jemermed.2022.10.009. Epub 2023 Jan 12. PMID 36641258